CLINICAL TRIAL: NCT04449926
Title: BCG and Plasma Amyloid in Non-Demented Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mindful Diagnostics and Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BCG-PANDA 01
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer Disease, Late Onset
Keywords: Alzheimer's disease; biomarker; BCG; plasma amyloid; peptides 42/40; heterologous effect; immune risk profile; CMV; HHV5; immunosenescence
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BCG Vaccinated (Experimental): Experimental: BCG Group FDA-approved BCG Tice strain, procured from Merck, will be used. The vaccine will be reconstituted according to the package insert. In brief, a vial containing ~1x10^8 CFU of lyophilized BCG will be reconstituted in 50 mL of saline. A single dose will consist of 0.1 mL (~2x10^5 CFU) will be administered by slow intradermal injection using a 25 gauge/ 0.5 mm syringe in the deltoid area. A follow up "booster" dose will be given one month after the initial dose.
  Interventions: Biological: Bacillus of Calmette and Guerin (BCG)

INTERVENTIONS:
Biological: Bacillus of Calmette and Guerin (BCG) — Prime and boost vaccination

SUMMARY:
BCG vaccination, the most widely used vaccination in the world, is used to reduce risk of tuberculosis infection; it is used for other mycobacterial infections as well, benefiting leprosy and Buruli ulcer. BCG has "heterologous" effects that aids in an array of non-mycobacterial and viral infections as well as bladder cancer. It is the heterologous effect, sometimes called the "off-target" effect that may offer benefit in Alzheimer's disease. Population studies and studies of adults receiving BCG show a lessened risk of Alzheimer's disease. The study will see if BCG vaccination will alter a plasma test for amyloid, a biomarker for cerebral amyloid.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is commonly regarded as Alzheimer's dementia. It is now understood that changes in the brain that result in late-onset AD dementia start years or even decades prior to clinical dementia. Biomarkers aid in diagnosing AD however, currently approved biomarkers have drawbacks as they are invasive and expensive. The two most commonly used biomarkers are amyloid PET scan and spinal tap for amyloid and tau. A new plasma amyloid test has received "Breakthrough Device Designation" from the US-FDA. As an investigational tool, this blood test for amyloid peptides 42/40 levels accurately predicts brain amyloidosis in cognitively normal individuals. In the past 100 years, four billion doses of BCG vaccination have been given for tuberculosis prevention. A favorable effect with BCG for non-tuberculous mycobacteria is also recognized in cervical lymphadeniits, leprosy and Buruli's ulcer. Recently, BCG has found favorable use in autoimmune diseases type 1 diabetes (T1D) and multiple sclerosis (MS); moreover, a protective role by BCG for Alzheimer's disease has been described. Adult exposure to BCG lessened the risk of AD by four-fold. This is an interventional pilot study to test 50 non-demented adults measuring their plasma amyloid 42/40 level prior to BCG prime/boost followed with the same plasma amyloid testing 9 months after vaccination. Sub-clinical CMV infection is felt to drive immune senescence and increase the risk of AD; we will test for CMV antibodies and we will measure lymphocyte phenotype prior to BCG and at study end to look for an immune-modulating effect on this indicator of immunosenescence.

ELIGIBILITY:
Inclusion Criteria:

* BCG naive
* Ability to read, understand and sign consent form

Exclusion Criteria:

* Known allergy to (components of) the BCG vaccine or serious adverse events to prior vaccine administration
* Known active or latent Mycobacterium tuberculosis or with another mycobacterial species. A history of - or a suspicion of M. tuberculosis infection.
* Fever (>38 C) within the past 24 hours.
* Suspicion of active viral or bacterial infection.
* Vaccination in the past 4 weeks or expected vaccination during the study period, independent of the type of vaccination.
* Severely immunocompromised subjects. This exclusion category comprises: a) subjects with known infection by the human immunodeficiency virus (HIV-1); b) neutropenic subjects with less than 500 neutrophils/mm3; c) subjects with solid organ transplantation; d) subjects with bone marrow transplantation; e) subjects under chemotherapy; f) subjects with primary immunodeficiency; g) severe lymphopenia with less than 400 lymphocytes/mm3; h) treatment with any anti-cytokine therapies. i) treatment with oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than 3 months, or probable use of oral or intravenous steroids in the following four weeks.
* Active solid or non-solid malignancy or lymphoma within the prior two years.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Amyloid | 9 months
  Level of Plasma Peptides 42/40 pre-BCG vaccination are compared with levels nine months post vaccination

SECONDARY OUTCOMES:
Change in Immune Risk Profile | nine months
  T-cell phenotype: CD4:CD8 ratios are measured pre-BCG vaccination and nine months post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Coad T Dow, M.D., Principal Investigator — Mindful Diagnostics and Therapeutics
Locations (1):
- Mindful Diagnostics and Therapeutics, Eau Claire, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schindler SE, Bollinger JG, Ovod V, Mawuenyega KG, Li Y, Gordon BA, Holtzman DM, Morris JC, Benzinger TLS, Xiong C, Fagan AM, Bateman RJ. High-precision plasma beta-amyloid 42/40 predicts current and future brain amyloidosis. Neurology. 2019 Oct 22;93(17):e1647-e1659. doi: 10.1212/WNL.0000000000008081. Epub 2019 Aug 1. PMID 31371569
- [Background] Gofrit ON, Klein BY, Cohen IR, Ben-Hur T, Greenblatt CL, Bercovier H. Bacillus Calmette-Guerin (BCG) therapy lowers the incidence of Alzheimer's disease in bladder cancer patients. PLoS One. 2019 Nov 7;14(11):e0224433. doi: 10.1371/journal.pone.0224433. eCollection 2019. PMID 31697701
- [Background] Gofrit ON, Bercovier H, Klein BY, Cohen IR, Ben-Hur T, Greenblatt CL. Can immunization with Bacillus Calmette-Guerin (BCG) protect against Alzheimer's disease? Med Hypotheses. 2019 Feb;123:95-97. doi: 10.1016/j.mehy.2019.01.007. Epub 2019 Jan 11. PMID 30696606
- [Background] Dow CT. Proposing BCG Vaccination for Mycobacterium avium ss. paratuberculosis (MAP) Associated Autoimmune Diseases. Microorganisms. 2020 Feb 5;8(2):212. doi: 10.3390/microorganisms8020212. PMID 32033287
- [Background] Lurain NS, Hanson BA, Martinson J, Leurgans SE, Landay AL, Bennett DA, Schneider JA. Virological and immunological characteristics of human cytomegalovirus infection associated with Alzheimer disease. J Infect Dis. 2013 Aug 15;208(4):564-72. doi: 10.1093/infdis/jit210. Epub 2013 May 9. PMID 23661800
- [Background] Westman G, Berglund D, Widen J, Ingelsson M, Korsgren O, Lannfelt L, Sehlin D, Lidehall AK, Eriksson BM. Increased inflammatory response in cytomegalovirus seropositive patients with Alzheimer's disease. PLoS One. 2014 May 7;9(5):e96779. doi: 10.1371/journal.pone.0096779. eCollection 2014. PMID 24804776
- [Background] Luz Correa B, Ornaghi AP, Cerutti Muller G, Engroff P, Pestana Lopes R, Gomes da Silva Filho I, Bosch JA, Bonorino C, Bauer ME. The inverted CD4:CD8 ratio is associated with cytomegalovirus, poor cognitive and functional states in older adults. Neuroimmunomodulation. 2014;21(4):206-12. doi: 10.1159/000356827. Epub 2014 Feb 6. PMID 24504177